CLINICAL TRIAL: NCT05773755
Title: Deep Brain Stimulation for Treatment Resistant Depression: Exploration of Local Field Potentials (LFPs) With the Medtronic Percept PC System
Brief Title: DBS for TRD With the Medtronic Percept PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Mayberg, MD (Other)
Responsible Party: Sponsor-Investigator, Helen Mayberg, MD, Professor, Neurology, Neurosurgery, Psychiatry and Neuroscience, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY-22-01731
Record Dates: First submitted 2023-02-21; First posted 2023-03-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: All participants will be implanted with the study device and receive open label, active DBS stimulation
Masking Description: N/A. This is open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Deep Brain Stimulation (DBS) for Treatment Resistant Depression (Experimental): Open label active Deep Brain Stimulation (DBS)
  Interventions: Device: Medtronic Percept PC DBS system

INTERVENTIONS:
Device: Medtronic Percept PC DBS system — Open label active Deep Brain Stimulation (DBS)

SUMMARY:
Of the estimated 30 million Americans who suffer from Major Depressive Disorder, approximately 10% are considered treatment resistant. Deep brain stimulation (DBS) to a region of the brain called the subcallosal cingulate (SCC) is an emerging strategy for treatment resistant depression (TRD), which involves placement of electrodes in a specific region of the brain and stimulating that area with electricity. This is believed to reset the brain network responsible for symptoms and results in a significant antidepressant response. A series of open-label studies have demonstrated sustained, long-term antidepressant effects in 40-60% of patients who received this treatment. A challenge to the effective dissemination of this fledgling treatment is the absence of biomarkers (objective, measureable indications of the state of the body and brain) to guide device placement and select stimulation parameters during follow-up care.

By using a DBS device called the Percept PC (Medtronic, Inc) which has the ability to both deliver stimulation to and record electrical signals directly from the brain, this study aims to identify changes in local field potentials (LFPs), specific electrical signals that are thought to represent how the brain communicates information from one region to another, to see how this relates to DBS parameter settings and patient depressive symptomatology. The goal of this study is to study LFPs before and during active DBS stimulation to identify changes that correlate with the antidepressant effects of SCC DBS.

The study team will recruit 10 patients with TRD and implant them with the Percept PC system. Participants will be asked to complete short questionnaires and collect LFP data twice daily for the first year of the study, as well as have weekly in person research procedures and assessments with the study team for up to one year. These include meetings with the study psychiatrist, psychologist, symptom ratings, and movement, voice, and video recordings. A brief discontinuation experiment will be conducted after 6 months of stimulation, in which the stimulation will be turned off and patterns of LFP changes will be recorded. The entire study is expected to last about 5 years, parcellated into several study phases. All participants are required to live in the New York metropolitan area for the first several months of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-70 years old.
* Ability to provide written informed consent.
* Primary psychiatric diagnosis of Major Depressive Disorder (MDD), either single episode or recurrent type, without psychotic features, currently experiencing a Major Depressive Episode (MDE), as diagnosed by Structured Clinical Interview for DSM IV-TR or DSM-5 (SCID-IV or SCID-5). Two independent psychiatrists will confirm the diagnosis, as well.
* Current depressive episode of at least two years duration OR a history of more than 3 lifetime depressive episodes.
* Minimum score at study entry of 20 on the 17-item Hamilton Depression Rating Scale
* Average pre-operative HDRS-17 score of 20 or greater (averaged over four weekly pre-surgical evaluations during the four weeks prior to surgery)
* A maximum Global Assessment of Functioning of 50 or less.
* Confirmed to have treatment-resistant depression (TRD). Treatment-resistance will be defined as failure to respond to at least four adequate antidepressant treatments (assessed with the Antidepressant Treatment History Form [ATHF-SF] and verified through medical records) during the current episode. Treatments which support study inclusion include antidepressive medications, certain augmentation agents, evidenced-based psychotherapy, and neuromodulation (ECT, transcranial magnetic stimulation (TMS)). For those patients who have not received ECT, patients may be considered eligible for study participation if they have received adequate trials of an SSRI, SNRI, augmentation agent (certain atypical antipsychotic medications, Lithium), and TMS and/or ketamine.
* ability comply with study and device management procedures.

Exclusion criteria:

* Other primary Axis I conditions
* Active suicidal ideation with intent, suicide attempt within the last six months, more than three suicide attempts within the last two years, or serious suicide risk as determined by the study psychiatrists
* Other primary neurological disorders or unstable medical illness
* Conditions requiring anticoagulant therapy which cannot be discontinued for the perioperative period, as required
* Pregnancy or plan to come pregnant during the study
* Contraindications for general anesthesia, neurosurgery, or an MRI scan
* Currently implanted with a cardiac pacemaker / defibrillator or other implanted electrical device which may interfere with DBS stimulator or the function of which may be impacted by its implantation.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HDRS) score | baseline and up to 1 year
  Response to intervention defined as a decrease in the HDRS-17 score of 50% or greater from the 4-week average pre-surgical baseline.
  Clinical remission will be defined as an HDRS-17 score ≤ 7. Partial response will be defined as a decrease in HDRS-17 >30% but less than 50%.
  Non-response will be defined as a <30% decrease in HDRS-17.
  The score for Hamilton Depression Rating Scale, 17 item version, ranges from 0-50, with a higher score indicating more severe depression.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | baseline and up to 1 year
  The MADRS consists of 10 items evaluating core symptoms of depression. Nine of the items are based upon patient report, and one is on the rater's observation during the rating interview. MADRS items are rated on a 0 to 6 continuum (0 = no abnormality, 6 = severe). Scores range from 0 to 60, with higher total scores indicating increased severity of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mayberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to helen.mayberg@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included in the URL field below).

REFERENCES:
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, Crowell AL, Garlow SJ, Rajendra JK, McIntyre CC, Gross RE, Mayberg HS. A connectomic approach for subcallosal cingulate deep brain stimulation surgery: prospective targeting in treatment-resistant depression. Mol Psychiatry. 2018 Apr;23(4):843-849. doi: 10.1038/mp.2017.59. Epub 2017 Apr 11. PMID 28397839
- [Background] Crowell AL, Riva-Posse P, Holtzheimer PE, Garlow SJ, Kelley ME, Gross RE, Denison L, Quinn S, Mayberg HS. Long-Term Outcomes of Subcallosal Cingulate Deep Brain Stimulation for Treatment-Resistant Depression. Am J Psychiatry. 2019 Nov 1;176(11):949-956. doi: 10.1176/appi.ajp.2019.18121427. Epub 2019 Oct 4. PMID 31581800
- [Background] Riva-Posse P, Crowell AL, Wright K, Waters AC, Choi K, Garlow SJ, Holtzheimer PE, Gross RE, Mayberg HS. Rapid Antidepressant Effects of Deep Brain Stimulation and Their Relation to Surgical Protocol. Biol Psychiatry. 2020 Oct 15;88(8):e37-e39. doi: 10.1016/j.biopsych.2020.03.017. Epub 2020 May 14. No abstract available. PMID 32418613
- [Background] Smart O, Choi KS, Riva-Posse P, Tiruvadi V, Rajendra J, Waters AC, Crowell AL, Edwards J, Gross RE, Mayberg HS. Initial Unilateral Exposure to Deep Brain Stimulation in Treatment-Resistant Depression Patients Alters Spectral Power in the Subcallosal Cingulate. Front Comput Neurosci. 2018 Jun 12;12:43. doi: 10.3389/fncom.2018.00043. eCollection 2018. PMID 29950982
- [Background] Waters AC, Veerakumar A, Choi KS, Howell B, Tiruvadi V, Bijanki KR, Crowell A, Riva-Posse P, Mayberg HS. Test-retest reliability of a stimulation-locked evoked response to deep brain stimulation in subcallosal cingulate for treatment resistant depression. Hum Brain Mapp. 2018 Dec;39(12):4844-4856. doi: 10.1002/hbm.24327. Epub 2018 Aug 18. PMID 30120851
- [Background] Veerakumar A, Tiruvadi V, Howell B, Waters AC, Crowell AL, Voytek B, Riva-Posse P, Denison L, Rajendra JK, Edwards JA, Bijanki KR, Choi KS, Mayberg HS. Field potential 1/f activity in the subcallosal cingulate region as a candidate signal for monitoring deep brain stimulation for treatment-resistant depression. J Neurophysiol. 2019 Sep 1;122(3):1023-1035. doi: 10.1152/jn.00875.2018. Epub 2019 Jul 17. PMID 31314668
- [Background] Howell B, Choi KS, Gunalan K, Rajendra J, Mayberg HS, McIntyre CC. Quantifying the axonal pathways directly stimulated in therapeutic subcallosal cingulate deep brain stimulation. Hum Brain Mapp. 2019 Feb 15;40(3):889-903. doi: 10.1002/hbm.24419. Epub 2018 Oct 11. PMID 30311317
- [Background] Smith EE, Choi KS, Veerakumar A, Obatusin M, Howell B, Smith AH, Tiruvadi V, Crowell AL, Riva-Posse P, Alagapan S, Rozell CJ, Mayberg HS, Waters AC. Time-frequency signatures evoked by single-pulse deep brain stimulation to the subcallosal cingulate. Front Hum Neurosci. 2022 Aug 18;16:939258. doi: 10.3389/fnhum.2022.939258. eCollection 2022. PMID 36061500
- [Background] Tiruvadi V, James S, Howell B, Obatusin M, Crowell A, Riva-Posse P, Gross RE, McIntyre CC, Mayberg HS, Butera R. Mitigating Mismatch Compression in Differential Local Field Potentials. IEEE Trans Neural Syst Rehabil Eng. 2023;31:68-77. doi: 10.1109/TNSRE.2022.3217469. Epub 2023 Jan 30. PMID 36288215
- [Background] Tiruvadi V, Choi KS, Gross RE, Butera R, Jirsa V, Mayberg H. Dynamic Oscillations Evoked by Subcallosal Cingulate Deep Brain Stimulation. Front Neurosci. 2022 Feb 23;16:768355. doi: 10.3389/fnins.2022.768355. eCollection 2022. PMID 35281513
- [Background] Harati S, Crowell A, Mayberg H, Nemati S. Depression Severity Classification from Speech Emotion. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:5763-5766. doi: 10.1109/EMBC.2018.8513610. PMID 30441645
- [Background] Harati S, Crowell A, Huang Y, Mayberg H, Nemati S. Classifying Depression Severity in Recovery From Major Depressive Disorder via Dynamic Facial Features. IEEE J Biomed Health Inform. 2020 Mar;24(3):815-824. doi: 10.1109/JBHI.2019.2930604. Epub 2019 Jul 23. PMID 31352356
- [Background] Harati S, Crowell A, Mayberg H, Nemati S. Addressing the Credit Assignment Problem in Treatment Outcome Prediction using Temporal Difference Learning. Pac Symp Biocomput. 2020;25:43-54. PMID 31797585
- [Background] Mazza A, Barucchi AM, Solimei GE, Viti M. [Clinical and immunological aspects of Lichen ruber planus]. Arch Stomatol (Napoli). 1988 Oct;29(4):657-66. Italian. PMID 3274606
- [Background] Riva-Posse P, Holtzheimer PE, Garlow SJ, Mayberg HS. Practical considerations in the development and refinement of subcallosal cingulate white matter deep brain stimulation for treatment-resistant depression. World Neurosurg. 2013 Sep-Oct;80(3-4):S27.e25-34. doi: 10.1016/j.wneu.2012.11.074. Epub 2012 Dec 13. PMID 23246630
- [Background] Crowell AL, Garlow SJ, Riva-Posse P, Mayberg HS. Characterizing the therapeutic response to deep brain stimulation for treatment-resistant depression: a single center long-term perspective. Front Integr Neurosci. 2015 Jun 15;9:41. doi: 10.3389/fnint.2015.00041. eCollection 2015. PMID 26124710
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, McIntyre CC, Gross RE, Chaturvedi A, Crowell AL, Garlow SJ, Rajendra JK, Mayberg HS. Defining critical white matter pathways mediating successful subcallosal cingulate deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2014 Dec 15;76(12):963-9. doi: 10.1016/j.biopsych.2014.03.029. Epub 2014 Apr 13. PMID 24832866
- [Background] Sendi MSE, Waters AC, Tiruvadi V, Riva-Posse P, Crowell A, Isbaine F, Gale JT, Choi KS, Gross RE, S Mayberg H, Mahmoudi B. Intraoperative neural signals predict rapid antidepressant effects of deep brain stimulation. Transl Psychiatry. 2021 Nov 3;11(1):551. doi: 10.1038/s41398-021-01669-0. PMID 34728599